CLINICAL TRIAL: NCT03324919
Title: Patient Centered Care Situation and Health-related Quality of Life of Patients From Non-urban Practice vs University Hospital With Diagnosis Psoriasis Vulgaris, Urticaria or Lupus Erythematodes
Brief Title: Patient Centered Care Situation and Health-related Quality of Life by Patients With Psoriasis, Urticaria or Lupus
Acronym: PUL
Status: Completed | Type: Observational
Sponsor: University Hospital Regensburg (Other)
Collaborators: University of Regensburg (Other)
Responsible Party: Principal Investigator, Tim Maisch, PD Dr., University Hospital Regensburg
Other Study IDs: UHRegensburg
Record Dates: First submitted 2016-03-14; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Quality of Life
Keywords: Psoriasis; Urticaria; Lupus erythematodes; qualtiy of life
MeSH Terms: conditions — Psoriasis; Urticaria

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Psoriasis, HRQL: Patients with a medical diagnosis of Psoriasis were enclosed.
  Interventions: Behavioral: HRQL
- Urticaria, HRQL: Patients with a medical diagnosis of Urticaria were enclosed.
  Interventions: Behavioral: HRQL
- Lupus erythematodes, HRQL: Patients with a medical diagnosis of Lupus were enclosed.
  Interventions: Behavioral: HRQL

INTERVENTIONS:
Behavioral: HRQL — Intervention of patient centered care situation and health-related quality of life of patients with Psoriasis, Urticaria or Lupus erythematodes from non-urban practices vs urban practises. Identification of relevant health-related quality of life parameters of these patients.
  Other Names: one-time survey

SUMMARY:
This study is based on a survey about the patient centered care situation and health-related quality of life of patients with diagnoses Psoriasis, Urtikaria or Lupus erythematodes. Detection of relevant parameters of quality of life by these patients serves for the detection of psychosocial burden of the mentioned skin diseases, thus gaining an increasing importance for prospective economic issues. This survey is a behaviorally based questionnaire for patients with the above diseases and addresses activities such as sleep and rest, mobility, recreation, home management, emotional behavior, social interaction, and the like.

DETAILED DESCRIPTION:
The care of patients with the above indications is based on a wide variety of available therapies. This study is based on a survey about the patient centered care situation and health-related quality of life of patients with diagnoses Psoriasis, Urtikaria or Lupus erythematodes. Therefore a cross-sectional survey will be done of patients with the above diseases from non-urban practices vs. urban practices (University Hospital). An adequate diagnosis and treatment of Psorisasis, Urticaria or Lupus erythematodes is often problematic due to the diverse and complex organ manifestations. However adequate diagnosis and appropriate treatments of these diseases is often conducted by various medical specialists in both outpatient and in-patient care. Lack of access and ability of the rural population to get an appropriate therapy may lead by these patients to false diagnosis or a therapeutic oversupply of an only symptom-oriented therapy. Furthermore the partly chronic character in the above mentioned diseases with recurrent symptoms, connected with prolonged itching periods and long-lasting treatments by these patients can lead to both emotional, mental stress and physical isolation. This situation does not only affect the health but also the overall quality of life of these patients. Therefore this study addresses several factors concerning the patient's perceived health status and to detect changes or differences in health status occurring between groups (patients from non-urban practices vs urban practices)

ELIGIBILITY:
Inclusion Criteria:

* Voluntary consent by written and oral explanation.
* Patients with the diseases Psoriasis, Urticaria or Lupus

Exclusion Criteria:

* Children and adolescents < 18 years
* pregnancy and breast feeding period of women
* History of abuse of alcohol, drugs or other substances, or factors that limit the ability to cooperate and compliance in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Psoriasis, Urticaria or Lupus erythematodes. History for the respective disease with the appropriate score classification by Guideline.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Investigation of patient centered care situation and health-related quality of life of patients with Psoriasis, Urtikaria and Lupus erythematosus | 24 months
  Detection of the quality of life score by these patients. Questionnaire administration and clinical documentation takes place when patients were present at the outpatient clinic of the Department of Dermatology, University Hospital Regensburg. Key inclusion criteria: diagnoses of psoriasis, urticaria or lupus erythematodes

SECONDARY OUTCOMES:
Identification of relevant health-related quality of life parameters of these patients | 24 months
  Questionnaire, that my medical care situation must be improved at all depending on my DLQI score. The DLQI-Questionnaire will be used.The questionnaires address skin-specific aspects as well as general aspects (activities of daily living, overall health-status) of quality of life.
Evalulation of the EQ5D-5L score of patients with Psoriasis, Urtikaria and Lupus erythematosus | 24 months
  EQ5D-5L Questionnaire and vas score, depending on the travel maximal distance accessing healthcare

CONTACTS AND LOCATIONS:
Overall Officials: Tim Maisch, PhD., Principal Investigator — University Hospital Regensburg, Department of Dermatology, Germany
Locations (1):
- University Hospital Regensburg, Regensburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bewley A, Burrage DM, Ersser SJ, Hansen M, Ward C. Identifying individual psychosocial and adherence support needs in patients with psoriasis: a multinational two-stage qualitative and quantitative study. J Eur Acad Dermatol Venereol. 2014 Jun;28(6):763-70. doi: 10.1111/jdv.12174. Epub 2013 May 13. PMID 23663069
- [Background] Kuhn A, Landmann A. The classification and diagnosis of cutaneous lupus erythematosus. J Autoimmun. 2014 Feb-Mar;48-49:14-9. doi: 10.1016/j.jaut.2014.01.021. Epub 2014 Jan 31. PMID 24486120
- [Background] Muller K, Karrer S, Apfelbacher C, Blome C, Berneburg M, Koller M. [Quality of life in dermatology. From measurement to practical implementation]. Hautarzt. 2015 Apr;66(4):287-96; quiz 297-8. doi: 10.1007/s00105-015-3599-8. German. PMID 25822586